CLINICAL TRIAL: NCT03956407
Title: Comparison Between Mechanisms Underlying Effects of Repetitive Peripheral Nerve Stimulation on Upper Limb Motor Performance in the Subacute and Chronic Phases After Stroke
Brief Title: Repetitive Nerve Stimulation to Improve Recovery After Stroke
Acronym: RESTORES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3019629
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: Rehabilitation; Neuromodulation; Peripheral stimulation; Motor function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: An amendment for performance of a minimization procedure in order to enhance the probability of comparable characteristics between the groups was approved. The researcher responsible for minimization is not involved in data collection or analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Suprathreshold, subacute stroke (Experimental): Repetitive peripheral sensory stimulation (RPSS) + Motor Training. Suprathreshold RPSS will be administered for 2 hours. After RPES, the patient will receive motor training.
  Interventions: Device: Suprathreshold repetitive peripheral sensory stimulation
- Subthreshold, subacute stroke (Other): Other: Subthreshold RPSS + Motor Training. Subthreshold RPSS will be administered for 2 hours. After RPSS, the patient will receive motor training
  Interventions: Device: Subthreshold repetitive sensory stimulation
- Suprathreshold, chronic stroke (Experimental): Repetitive peripheral sensory stimulation (RPSS) + Motor Training. Suprathreshold RPSS will be administered for 2 hours. After RPSS, the patient will receive motor training.
  Interventions: Device: Suprathreshold repetitive peripheral sensory stimulation
- Subthreshold, chronic stroke (Other): Other: Subthreshold RPSS + Motor Training. RPSS will be administered for 2 hours. After RPSS, the patient will receive motor training
  Interventions: Device: Subthreshold repetitive sensory stimulation

INTERVENTIONS:
Device: Suprathreshold repetitive peripheral sensory stimulation — Suprathreshold repetitive peripheral sensory stimulation will be applied to the median nerve of the affected forearm with surface electrodes. The stimulator will be set to deliver bursts of 10 Hz stimulation at 50% duty cycle (500 ms on and off). For suprathreshold stimulation, intensities will be set at the highest intensity able to induce sensory paraesthesias without overt muscle contraction or pain, and adjusted if required.
  Arms: Suprathreshold, chronic stroke; Suprathreshold, subacute stroke
Device: Subthreshold repetitive sensory stimulation — Subthreshold repetitive sensory stimulation will be applied to the median nerve of the affected forearm with surface electrodes. The stimulator will be set to deliver bursts of 10 Hz stimulation at 50% duty cycle (500 ms on and off). For subthreshold stimulation, intensities will be set at 10mv - 15mv lower than de lowest intensity able to induce sensory paraesthesias, and adjusted if required.
  Arms: Subthreshold, chronic stroke; Subthreshold, subacute stroke

SUMMARY:
Upper limb paresis is the most common type of post-stroke neurological impairment and a major cause of functional disability. Repetitive peripheral sensory stimulation (RPSS) is a novel strategy to improve upper limb motor performance in the post-stroke chronic phase but its effects in the subacute phase are still poorly understood. The objectives of this study are to compare the effects of RPSS on motor performance of the upper limb in the subacute and chronic phases of stroke, and to identify the mechanisms underlying this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke confirmed by computed tomography or magnetic resonance imaging, between 7 days - 3 months before enrollment (subacute phase), and at least 6 months (chronic phase).
* Ability to perform at least 4 of 7 tasks performed in daily life that is part of the Jebsen-Taylor Test

Exclusion Criteria:

* Anesthesia of the paretic hand.
* Lesions affecting the motor cortex (hand area).
* Lesions affecting cerebellum, or cerebellar pathways in the brainstem.
* Severe spasticity at the paretic elbow, fist or fingers, defined with a score larger than 3 on the Modified Ashworth Scale.
* Neurological diseases such as Parkinson disease or chronic uncontrolled chronic disease such as cancer or cardiac insufficiency.
* Elbow pain or join deformity in the paretic limb.
* Pregnancy.
* Uncontrolled psychiatric disease.
* Aphasia or severe cognitive deficit.
* Inability to provide consent.
* Inability to attend the experimental sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Jebsen-Taylor Test | Immediately after one session of intervention
  Test of upper limb dexterity

SECONDARY OUTCOMES:
Change in lateral pinch strength | Immediately after one session of intervention
  Pinch strength measured with dynamometer
Change in gamma-aminobutyric acid levels in primary motor cortex | Immediately after one session of intervention
  Gamma-aminobutyric acid levels measured with magnetic resonance imaging spectroscopy
Change in brain perfusion | Immediately after one session of intervention
  Brain perfusion measured with magnetic resonance imaging - arterial spin labeling
Change in grasp strength | Immediately after one session of intervention
  Grasp strength measured with dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital São Rafael, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kroth JB, Handfas B, Rodrigues G, Zepeda F, Oliveira MA, Wang DJJ, de Azevedo Neto RM, Silva GS, Amaro E Jr, Sorinola IO, Conforto AB. Effects of Repetitive Peripheral Sensory Stimulation in the Subacute and Chronic Phases After Stroke: Study Protocol for a Pilot Randomized Trial. Front Neurol. 2022 Feb 16;13:779128. doi: 10.3389/fneur.2022.779128. eCollection 2022. PMID 35250807